CLINICAL TRIAL: NCT04005196
Title: EEG Phase SynchrOny, Sedation and Delirium in the CVICU - The SOS Study
Brief Title: EEG Phase Synchrony, Sedation and Delirium in the CVICU
Acronym: SOS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Toronto (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, M. Elizabeth Wilcox, Assistant Professor, University of Toronto
Other Study IDs: 17-6037
Record Dates: First submitted 2019-06-30; First posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-07

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium | interventions — Electroencephalography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: EEG — Data recording will continue up until a maximum of 120 hours after emergence from sedation or at CVICU discharge. This study period is informed by baseline data from our institution where the median duration of delirium following emergence from coma was 2 days, allowing sufficient time to capture transitions from coma to wakefulness with and without delirium. EEG recordings will be divided in to epochs corresponding to coma, wakefulness, and delirium if present.

SUMMARY:
EEG phase synchrony and variability has had limited investigation during transition from coma to wakefulness in response to sedation and analgesia. Studying changes in phase synchrony and variability during and after sedative-induced coma is an exciting opportunity to better understand EEG changes during transitions in states of arousal. It is expected that consciousness should be higher in entropy and greater in complexity in the number of configurations of pairwise connections as compared to sedative-induced coma. If sufficiently sensitive, it may be possible to identify states of lower entropy and fewer configurations when patient are aroused but with altered sensorium (e.g. delirium).

DETAILED DESCRIPTION:
Aim 1: To quantify EEG phase synchrony changes, both globally and locally by brain region, during emergence from medically induced coma required for performance of a cardiovascular related operation (deep sedation defined as a Riker Sedation-Agitation Scale [SAS] of 1-2).

Hypothesis: The global R-index will be increased above baseline at multiple frequency bandwidths and the magnitude of R-index will correlate with the sedative dosage (as a crude measure of depth). The rate of fluctuations of the R-index will decrease with deeper sedation.

Aim 2: To compare the magnitude of the EEG phase synchrony globally and locally in patients emerging from coma; a patient's pre-anesthesia phase will serve as a control.

Hypothesis: Fluctuations in R-index will vary; fluctuations will be greater in awake adults as compared to while comatose or emerging from coma.

Aim 3: To determine EEG phase synchrony changes in patients with and without delirium during their CVICU stay.

Hypothesis: Lower scores of R-index consistent with increased phase synchrony and lower spatio-temporal variability will be seen while delirious as compared to days when patients are not delirious.

ELIGIBILITY:
Inclusion criteria:

* Age 30 - 65 years
* Scheduled for first-time CABG or single valve replacement

Exclusion criteria:

* Previous stroke
* Severe pre-existing cognitive impairment (TICS score < 24)

Ages: 30 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Population: Adults aged 30 - 65 years, invasively mechanically ventilated for a first-time CABG or single valve replacement surgery; Exposure: R-index measured at different states of consciousness (awake, emerging from comatosed state, and transitional states between) after standardized induction with opioid and benzodiazepine with or without propofol; postoperative sedation in CVICU with propofol or other; Outcome: Delirium as measured by the Confusion Assessment Method-ICU (CAM-ICU).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Electroencephalography (EEG) | Until ICU discharge; to a maximum 21 days
  R-Index -- phase synchrony

SECONDARY OUTCOMES:
CAM-ICU | Until ICU discharge; to a maximum 21 days
  q6 hours while in the ICU: delirium screen instrument

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network - Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided